CLINICAL TRIAL: NCT06465953
Title: A Phase 3, Multicenter, Open Label, Randomized, Non-comparative Two-arm Study of Ivosidenib (IVO) Monotherapy and Azacitidine (AZA) Monotherapy in Adult Patients With Hypomethylating Agent (HMA) Naive Myelodysplastic Syndromes (MDS) With an Isocitrate Dehydrogenase-1 (IDH1) Mutation (PyramIDH Study)
Brief Title: Ivosidenib (IVO) Monotherapy and Azacitidine (AZA) Monotherapy in Patients With Hypomethylating Agent (HMA) Naive Myelodysplastic Syndromes (MDS) With an IDH1 Mutation
Acronym: PyramIDH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: Servier Bio-Innovation LLC (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S095031-178; 2023-510155-37 (EudraCT Number)
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hypomethylating Agent (HMA) Naive Myelodysplastic Syndromes (MDS); Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — ivosidenib; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivosidenib monotherapy (Experimental)
  Interventions: Drug: Ivosidenib
- Azacitidine monotherapy (Experimental)
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Ivosidenib — Two 250 mg tablets, totaling 500 mg, administered orally once daily until disease relapse or progression, unacceptable toxicity, confirmed pregnancy, undergoing HSCT, death, withdrawal of consent, lost to follow-up, or Sponsor ending the study, whichever occurs first.
  Arms: Ivosidenib monotherapy
Drug: Azacitidine — Azacitidine 75mg/m^2/day administered by subcutaneous (SC) or intravenous (IV) injection for 1 week (7 days) of each 4-week (28 day) treatment cycle until disease relapse or progression, unacceptable toxicity, confirmed pregnancy, undergoing HSCT, death, withdrawal of consent, lost to follow-up, or Sponsor ending the study, whichever occurs first.
  Arms: Azacitidine monotherapy

SUMMARY:
This study will enroll participants with myelodysplastic syndromes (MDS) with an Isocitrate dehydrogenase protein, 1 (IDH1) mutation, who have not received treatment with a hypomethylating agent previously. Participants will be randomized to receive either ivosidenib (IVO) alone or azacitidine (AZA) alone. IVO will be administered daily throughout the 28-day treatment cycle and AZA will be administered for the first 7 days of each 28-day cycle. Study visits will be conducted every week during Cycle 1 (Days 1, 8, 15, and 22), and Day 1 of each cycle thereafter. After the last dose of treatment, participants will attend an safety follow-up visit and participants will be followed to assess overall survival. Study visits may include a bone marrow aspirate, physical exam, echocardiogram (ECHO), electrocardiogram (ECG), blood and urine analysis, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HMA naive IDH1 R132 mutated MDS defined according to WHO criteria (5th edition):
* Moderate high, high and very high-risk MDS per IPSS-M score will be eligible regardless of blood counts and with blast counts 0-19%.
* Low and moderate low-risk MDS per IPSS-M score must:
* Have cytopenias related to MDS, defined as: <100 platelets/microliter, or absolute neutrophil count (ANC) <1000/mm3, or hemoglobin <10g/dL AND
* Have a blast count between 5-19% AND
* Be eligible for HMA therapy (very low risk participants are to be excluded)
* Locally or centrally confirmed IDH1 R132 C/G/H/L/S mutation

Exclusion Criteria:

* Received prior anticancer/disease modifying treatment for MDS (including HMA's, cytotoxic chemotherapy, investigational agents, bcl-2 inhibitor based-regimens, hematopoietic stem cell transplant (HSCT), IDH1 inhibitors). For LR-MDS patients, prior treatment with growth factors, luspatercept, lenalidomide, and imetelstat are allowed.
* >20% blasts by morphology or immunohistochemistry on screening bone marrow aspirate/biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving CR and PR by 4 months | Through 4 months after starting treatment
  Complete remission (CR) or Partial remission (PR) as per International Working Group (IWG) 2006 criteria

SECONDARY OUTCOMES:
Overall Response (OR) rate per IWG 2023 criteria | Through the end of the study (approximately 4 years)
  Defined as CR (or CR equivalent) + PR + CRL + CRh + hematological improvement (HI)
Event-free survival (EFS) | Through the end of the study (approximately 4 years)
  Defined as the date of randomization to the date of first documented confirmed relapse /progression /death, whichever occurs first
Overall Survival (OS) | Through the end of the study (approximately 4 years)
  Defined as the time from randomization to the date of death due to any cause. Participants who are alive at the analysis cutoff date will be censored at the date they were last known to be alive.
Duration of CR and PR | Through the end of the study (approximately 4 years)
  Among participants who achieved CR+PR per IWG 2006 criteria
Time to CR and PR | Through the end of the study (approximately 4 years)
  Defined as time from the date of the randomization to the date of CR+PR, among participants who achieve CR+PR based on IWG 2006 Response Criteria
Acute myeloid leukemia (AML) transformation rate | Through the end of the study (approximately 4 years)
Time to transfusion independence (TTTI) | Through the end of the study (approximately 4 years)
  Defined as time from date of randomization to date transfusion independence (TI) is first observed (Day 1 of a ≥ 56 days period without a transfusion), among participants who are baseline transfusion dependent and have achieved post-baseline TI. In the event a participant had more than one ≥ 56-day period, which met TI criteria, the earliest period will be used in analysis.
Duration of transfusion independence (DOTI) | Through the end of the study (approximately 4 years)
  Among participants who have achieved post-baseline TI, DOTI will be calculated as the time from the date TI is first observed (Day 1 of a ≥ 56-day period without a transfusion) until the day before the participants had a subsequent transfusion.
Transfusion independence rate | Through the end of the study (approximately 4 years)
Change from baseline in Quality of life (QOL) based on the QUALMS score | Through the Event Free Survival Follow up (approximately 4 years)
  Quality of Life in Myelodysplasia Scale (QUALMS) scores range from 0 to 100, with a higher score representing a better QOL.
Change from baseline in health economic outcomes measures based on EQ-5D-5L score | Through the Event Free Survival Follow up (approximately 4 years)
  Health economic outcomes measures as assessed by the 5-level EuroQol five dimensions questionnaire (EQ-5D-5L) scores range from 5 to 25 with a higher number representing a worse health status.
Number of participants who proceed to hematopoietic stem cell transplantation (HSCT) | Through the end of the study (approximately 4 years)
Ivosidenib plasma concentrations | Through Cycle 22 (each cycle is 28 days)
  For participants receiving ivosidenib monotherapy
2-HG plasma concentrations | Through Cycle 22 (each cycle is 28 days)
  For participants receiving ivosidenib monotherapy
Number of participants achieving CR and PR by 6 months as per IWG 2006 criteria | Through 6 months after starting treatment
Number of participants achieving CR and PR by 6 months as per IWG 2023 criteria | Through 6 months after starting treatment
Number of participants achieving CR and PR by 4 months as per IWG 2023 criteria | Through 4 months after starting treatment
Number of adverse events (AEs) and serious adverse events (SAEs) | Through the Safety Follow-up Visit (30-35 days after discontinuation of treatment)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (9):
  - Presbyterian / St. Luke'S Medical Center, Denver, Colorado
  - University of Chicago, Duchossois Center for Advanced Medicine (DCAM), Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - MSKCC, New York, New York
  - Unc Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - University of Texas UT Southwestern Comprehensive Cancer Center, Dallas, Texas
  - MD Anderson Cancer Centre, Houston, Texas
- Australia (6):
  - Royal Adelaide Hospital, Adelaide
  - Monash Health, Clayton
  - Northern Health, Epping
  - Liverpool Hospital, Liverpool
  - Sir Charles Gairdner Hospital, Nedlands
  - Calvary Mater Newcastle, Waratah
- Brazil (8):
  - Liga Paranaense de Combate ao Câncer - Hospital Erasto Gaertner, Curitiba
  - Centro de Pesquisa Clínica - Hospital Nove de Julho, São Paulo
  - Real E Benemérita Associação Portuguesa de São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Casa de Saúde Santa Marcelina, São Paulo
  - Centro de Pesquisas Clínicas da Fundação Doutor Amaral Carvalho, São Paulo
  - Instituto Nacional do Câncer, São Paulo
- France (6):
  - Chu Nantes-Hotel Dieu, Nantes
  - Chu de Nice - Hôpital L'Archet 1, Nice
  - Hopital Saint Louis, Paris
  - Chu Bordeaux, Hopital Du Haut Leveque, Pessac
  - Institut Universitaire Du Cancer Toulouse-Oncopole, Toulouse
  - Chu Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Universitatsklinikum Dresden Carl Gustav Carus, Dresden
  - Marien Hospital Duesseldorf, Düsseldorf
  - Universitaetsmedizin Goettingen (Umg), Göttingen
  - Universitaetsklinikum Leipzig, Leipzig
  - Tum Klinikum Rechts Der Isar, Munich
- Italy (7):
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Istituto Di Ematologia "Lorenzo E Ariosto Seragnoli" - Policlinico Di S. Orsola, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Humanitas Research Hospital (Istituto Clinico Humanitas), Milan
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Dipartimento Di Biomedicina E Prevenzione - Universita Degli Studi Di Roma "Tor Vergata", Roma
  - Azienda Ospedaliera Universitaria Citta Della Salute E Della Scienza Di Torino - Presidio Molinette, Torino
- Japan (6):
  - University of Fukui Hospital, Yoshida-gun, Eiheiji-cho 670-8540 Himeji
  - Kyushu University Hospital, Higashi-ku, Fukuoka-city, Fukuoka
  - Japanese Red Cross Society Himeji Hospital, Himeji-city, Hyogo
  - Tokai University Hospital, Isehara-city, Kanagawa
  - Japanese Red Cross Musashino Hospital, Musashino-city, Tokyo
  - Kitasato University Hospital, Sagamihara
- Netherlands (2):
  - Umc Amsterdam - Vumc, Amsterdam
  - Umc Groningen, Groningen
- Spain (7):
  - Institut Catala D' Oncologia, Badalona
  - H. Valle de Hebron, Barcelona
  - Clinica Universitaria de Navarra (Madrid), Madrid
  - Clinica Universitaria de Navarra (Pamplona), Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen de La Macarena, Seville
  - H. Universitario La Fe, Valencia
- United Kingdom (6):
  - Western General Hospital, Edinburgh
  - St James' University Hospital, Leeds
  - University College London Hospital, London
  - Kings College Hospital, London
  - Churchill Hospital, Oxford
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data. Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/